CLINICAL TRIAL: NCT03312296
Title: Definite Stent Thrombosis in Comatose Out of Hospital Cardiac Arrest Survivors Treated With Percutaneous Coronary Intervention and Hypothermia
Brief Title: Definite Stent Thrombosis in Comatose Out of Hospital Cardiac Arrest Survivors
Acronym: ST OHCA
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Marko Noc, Marko Noc, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: Stent thrombosis OHCA
Record Dates: First submitted 2017-10-12; First posted 2017-10-17 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Out of Hospital Cardiac Arrest; Stent Thrombosis; Drug Eluting Stent; Therapeutic Hypothermia
Keywords: Stent Thrombosis
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Reliable data on stent thrombosis (ST) in comatose out of hospital cardiac arrest (OHCA) survivors is lacking. In comatose OHCA survivors suspicion of ST can be made with precise clinical monitoring of the patient with definite confirmation being possible only by coronary angiography or autopsy of deceased patients. However in addition to definite ST which can be confirmed using current protocols, additional ST which are clinically silent are plausible. These could be identified only by systematic coronary angiography of all OHCA survivors or by autopsy of deceased patients. Collectively with definite ST confirmed by coronary angiography upon clinical suspicion the incidence of all forms of ST in survivors of OHCA treated with PCI and hypothermia could be obtained.

Consecutive comatose survivors of OHCA treated with percutaneous coronary intervention (PCI) and hypothermia will be included. All study participants will receive treatment per our established clinical protocol and will be followed for 10 days. In all patients in whom clinical suspicion of ST will be made immediate coronary angiography and if necessary PCI will be carried out. In all patients that will die in the observed period of 10 days autopsy will be performed. Survivors however will have an additional control coronary angiography on 10th day after admission, to assess presence of clinically silent ST.

We expect that the incidence of true definitive ST in comatose OHCA survivors treated with urgent PCI with stenting and hypothermia is greater than one, which is confirmed on the basis of clinical suspicion by angiography or later with autopsy.

ELIGIBILITY:
Inclusion Criteria:

* Comatose out-of-hospital cardiac arrest survivors admitted to University Medical Centre Ljubljana
* Treated with primary PCI with stenting
* Treated with therapeutic hypothermia.

Exclusion Criteria:

* Younger than 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Comatose survivors after out-of-hospital cardiac arrest admitted to University Medical Centre Ljubljana
Sampling Method: Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2021-08 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Incidence of definite early ST until day 10 | 10 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noc M, Fajadet J, Lassen JF, Kala P, MacCarthy P, Olivecrona GK, Windecker S, Spaulding C; European Association for Percutaneous Cardiovascular Interventions (EAPCI); Stent for Life (SFL) Group. Invasive coronary treatment strategies for out-of-hospital cardiac arrest: a consensus statement from the European association for percutaneous cardiovascular interventions (EAPCI)/stent for life (SFL) groups. EuroIntervention. 2014 May;10(1):31-7. doi: 10.4244/EIJV10I1A7. PMID 24832635
- [Background] Steblovnik K, Blinc A, Bozic-Mijovski M, Kranjec I, Melkic E, Noc M. Platelet reactivity in comatose survivors of cardiac arrest undergoing percutaneous coronary intervention and hypothermia. EuroIntervention. 2015 Apr;10(12):1418-24. doi: 10.4244/EIJY14M05_02. PMID 24800722
- [Background] Joffre J, Varenne O, Bougouin W, Rosencher J, Mira JP, Cariou A. Stent thrombosis: an increased adverse event after angioplasty following resuscitated cardiac arrest. Resuscitation. 2014 Jun;85(6):769-73. doi: 10.1016/j.resuscitation.2014.02.013. Epub 2014 Feb 23. PMID 24572484
- [Background] Knafelj R, Radsel P, Ploj T, Noc M. Primary percutaneous coronary intervention and mild induced hypothermia in comatose survivors of ventricular fibrillation with ST-elevation acute myocardial infarction. Resuscitation. 2007 Aug;74(2):227-34. doi: 10.1016/j.resuscitation.2007.01.016. Epub 2007 Mar 23. PMID 17383070
- [Background] Cutlip DE, Windecker S, Mehran R, Boam A, Cohen DJ, van Es GA, Steg PG, Morel MA, Mauri L, Vranckx P, McFadden E, Lansky A, Hamon M, Krucoff MW, Serruys PW; Academic Research Consortium. Clinical end points in coronary stent trials: a case for standardized definitions. Circulation. 2007 May 1;115(17):2344-51. doi: 10.1161/CIRCULATIONAHA.106.685313. PMID 17470709
- [Background] Bednar F, Kroupa J, Ondrakova M, Osmancik P, Kopa M, Motovska Z. Antiplatelet efficacy of P2Y12 inhibitors (prasugrel, ticagrelor, clopidogrel) in patients treated with mild therapeutic hypothermia after cardiac arrest due to acute myocardial infarction. J Thromb Thrombolysis. 2016 May;41(4):549-55. doi: 10.1007/s11239-015-1274-7. PMID 26340851
- [Background] Rosillo SO, Lopez-de-Sa E, Iniesta AM, de Torres F, del Prado S, Rey JR, Armada E, Moreno R, Lopez-Sendon JL. Is therapeutic hypothermia a risk factor for stent thrombosis? J Am Coll Cardiol. 2014 Mar 11;63(9):939-40. doi: 10.1016/j.jacc.2013.09.028. Epub 2013 Oct 16. No abstract available. PMID 24140665